CLINICAL TRIAL: NCT06622317
Title: Abdominal Aortic Junction Tourniquet (AAJT-S) for Non-compressible Torso Haemorrhage: a Prospective Observational Pilot Study
Brief Title: Abdominal Aortic Junction Tourniquet (AAJT-S) for Non-compressible Torso Haemorrhage
Status: Recruiting | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: 1063/2024
Record Dates: First submitted 2024-09-10; First posted 2024-10-02 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Exanguination; NCTH; Polytrauma
Keywords: NCTH; aortic occlusion; exanguniation
MeSH Terms: conditions — Multiple Trauma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

SUMMARY:
This study seeks to evaluate the feasibility of a Abdominal Aortic Balloon Occlusion of the Aorta (AAJT-S) in exanguinating trauma patients with non-compressible truncal haemorrhage in the emergency room and the pre-hospital setting.

DETAILED DESCRIPTION:
The study is designed as a prospective observational study to accomapany the impementation of this device in clinical routine. However, the device has already been used in the emergency room and AAJT-S application is no study specific intervention.

ELIGIBILITY:
Inclusion Criteria:

* aged, or believed to be aged, 18 years or above,
* confirmed or suspected life-threatening lower body trauma (i.e. signs of inadequate perfusion of tissues, tachycardia, hypotension, suspected blood loss)
* is thought to benefit from trauma resuscitation with AAJT-S or REBOA zone III

Exclusion Criteria:

* suspected additional bleeding source proximal to the umbilicus, or
* known or suspected pregnancy at presentation, or
* known abdominal aortic aneurysm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all patients meeting the eligibility criteria that are being transported to the rescucitation room of the Medical University of Graz
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2026-09-17 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
effective placement of the device | 1 hour
  cessation of bloodflow distal to the device

SECONDARY OUTCOMES:
30-day mortality | 30 days
  in-hospital
Complications | 90 days
  Occurrence of complications of device application
Heart rate | 1 hour
  Improvement (reduction) in beats/minute
Base excess | 1hour
  Improvement (reduction) in mmol/l
Blood pressure (systolic and diastolic) | 1 hour
  Improvement in mmHg

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Graz, Graz, Styria, Austria

IPD SHARING:
Plan to Share IPD: Undecided